CLINICAL TRIAL: NCT05694611
Title: Contrast Enhanced Ultrasound and Elastography of the Preterm Brain
Brief Title: Preterm Neonates Brain Ultrasound With CEUS and Elastography
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The recruitment conditions could'n be met, because the clinically based treatment plans were changed before the beginning of recruitment and the ex-preemies didn't have venous access at the time of examinations.
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Tiina Laurikainen, Principal Investigator, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TL16102021.1
Record Dates: First submitted 2022-12-05; First posted 2023-01-23 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth | interventions — Sulfur Hexafluoride; contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preterm neonates (Experimental): Diagnostic Test: Brain ultrasound, brain contrast enhanced ultrasound, brain ultrasound elastography To study brain perfusion with brain ultrasound, contrast enhanced ultrasound of the brain and ultrasound-guided shear-wave elastography Drug: Sulfur Hexafluoride To evaluate brain perfusion at term in infants born prematurely
  Other Names:
  • SonoVue
  Interventions: Diagnostic Test: Brain contrast enhanced ultrasound, brain ultrasound elastography; Drug: Sulfur Hexafluoride

INTERVENTIONS:
Diagnostic Test: Brain contrast enhanced ultrasound, brain ultrasound elastography — To study brain perfusion with brain ultrasound, contrast enhanced ultrasound of the brain and ultrasound-guided shear-wave elastography
Drug: Sulfur Hexafluoride — To evaluate the differences in brain perfusion and elasticity studied by CEUS and shear-wave elastography, comparing term neonates with and without MRI verified brain pathologies and to compare the ultrasound CEUS and elastography data to MRI.
  Other Names: SonoVue

SUMMARY:
The aim of the study is to investigate levels of brain perfusion and elasticity in preterm neonates when they reach the estimated due date and to compare the data with magnetic resonance imaging at term. Contrast enhanced ultrasound (sulphur hexafluoride) and ultrasound-assisted elastography will be used to evaluate the state of brain perfusion with ultrasound. Different appropriate imaging sequences will be used regarding MRI, including asl-perfusion. Neonates recruited from the Neonatal Intensive Care Unit (NICU) of Turku University Hospital will be recruited.

DETAILED DESCRIPTION:
SonoVue (sulphur hexafluoride) is a contrast agent composed of micro bubbles. It increases echogenicity of the ultrasound thus enhancing the visualisation of vessels and giving better insights into tissue perfusion. The use of sulphur hexafluoride has been approved by FDA and it has been in off-label use in Europe for years. SonoVue is thought to be especially useful for children, because it can enhance the diagnostic capabilities of ultrasound and the examination can be performed without radiation or sedation.

Elastography is a method to investigate the elasticity of a tissue by tracking the shear waves generated by the ultrasound beam. Also this method has been used in Europe and America for years.

The aim of this study is to examine cerebral hemodynamics in preterm neonates reaching term age, using ultrasound of the brain, contrast enhanced ultrasound (CEUS) and ultrasound-guided shear-wave elastography (US-SWE). The brain ultrasound, CEUS and US-SWE to preterm babies is planned to take place while having a clinically appointed brain magnetic resonance imaging at about term. Total recruitment for the study is 100 infants in total. The recruitment period will be up to seven years if needed.

The injections of SonoVue will be administered through pre-existing venous cannulas. The examination will be done in addition to the MR-imaging, after the parental consent has been given. The ultrasound examination altogether is estimated to take about 20 minutes per day. Safety monitoring period is conducted after the injection. CEUS data will be analysed with proper software. US-SWE will be measured repeatedly on both brain hemispheres and on different areas to validate the measurements. Ultrasound data will be evaluated comparing preterm neonates with and without MRI-proven brain pathology and comparing the ultrasound-achieved data to magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates attending brain MR-imaging at term

Exclusion Criteria:

* Pre-known genetic disease
* Difficult congenital malformations that need surgical treatment
* Central nervous system tumors
* Weight less than 2,5 kg during examination
* Medical history of SonoVue hypersensitivity
* Uncontrolled systemic hypertension
* Systolic pulmonary artery pressure > 90 mmHg
* Unstable cardiovascular state

Ages: 3 Weeks to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative assessment of neonatal brain perfusion using calculated time-intensity curve of enhancement in brain CEUS at term | 1 day
  Quantitative analysis will be executed from a time-intensity curve generated from a region of interest and from left and right talami. Wash-in slope and wash-out slope (measured in echo power units per second) will be measured and compared on healthy versus diseased preterm neonates at term.
Quantitative assessment of neonatal brain peak enhancement using calculated time-intensity curve of enhancement in brain CEUS at term | 1 day
  Quantitative analysis will be executed from a time-intensity curve generated from a region of interest and from left and right talami. Peak enhancement will be measured as maximum echo power on time-intensity curve.
Quantitative assessment of neonatal brain perfusion time to peak using calculated time-intensity curve of enhancement in brain CEUS at term | 1 day
  Quantitative analysis will be executed from a time-intensity curve generated from a region of interest and from left and right talami. Time to peak will be measured in seconds in time-intensity curve.
Quantitative assessment of neonatal brain perfusion volume using calculated time-intensity curve of enhancement in brain CEUS at term | 1 day
  Quantitative analysis will be executed from a time-intensity curve generated from a region of interest and from left and right talami. Area under the curve reporting total enhancement volume from time-intensity curve.

SECONDARY OUTCOMES:
Neonatal brain perfusion assessed with time-intensity curves of contrast enhanced ultrasound compared with brain magnetic resonance asl perfusion imaging | 1 day
  Time-intensity curves of CEUS and MRI ASL-perfusion studies will be performed comparing time to peak, peak enhancement, wash-in and wash-out curves and mean transit times on different imaging methods. Assessment will be done in correlation with clinical information.
Qualitative assessment of neonatal brain elasticity using ultrasound-guided shear wave elastography | 1 day
  Quantitative analysis of repeated US-SWE measurements on both hemispheres of thalami and areas of interest estimated by brain ultrasound and elastography. Tissue elasticity will be reported in kilopascals, comparing the findings of thalami and regions of interest on the left and on the right.

CONTACTS AND LOCATIONS:
Overall Officials: Tiina Laurikainen, Principal Investigator — Turku University Hospital; Riitta Parkkola, Study Director — Turku University Hospital; Vilhelmiina Parikka, Study Chair — Turku University Hospital; Jussi Hirvonen, Study Chair — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Southwestern Finland, Finland

IPD SHARING:
Plan to Share IPD: No